CLINICAL TRIAL: NCT04821297
Title: An Innovative and Linguistically-Tailored Mobile Intervention to Improve Follow-Up for Abnormal Pap Test Results: CervixChat
Brief Title: Linguistically-Tailored Mobile Intervention for the Improvement of Follow Up for Abnormal Pap Test Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20D.1271; JT 16196 (Other: JeffTrial Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Health Promotion; Educational Status; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (message) (Experimental): Patients receive text messages for 1-2 months before scheduled appointment. Patients also complete a survey at baseline and after standard of care colposcopy and an interview after standard of care colposcopy.
  Interventions: Other: Health Promotion and Education; Other: Survey Administration; Other: Interview

INTERVENTIONS:
Other: Health Promotion and Education — Receive messages
Other: Survey Administration — Complete survey
Other: Interview — Participate in an interview

SUMMARY:
This clinical trial evaluates the feasibility of a linguistically-tailored mobile intervention, called CervixChat in improving the follow-up of patients with abnormal Papanicolaou (pap) test results. A text messaging program, such as CervixChat may support patients who need a colposcopy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of CervixChat intervention in a mix method design, through participants consent rate and the study completion rate.

SECONDARY OBJECTIVE:

I. To evaluate the acceptability of CervixChat intervention using a validated Likert-scale participant satisfaction questionnaire, as well as participant's interview data.

EXPLORATORY OBJECTIVE:

I. To evaluate the preliminary impact of CervixChat intervention, by comparing the colposcopy appointment adherence rate in the study cohort against a 1:1 matched control sample selected based on matching age, race and ethnicity, from participants at Jefferson Obstetrics and Gynecology (Ob-Gyn) department scheduled for a colposcopy in 2019.

OUTLINE:

Patients receive text messages for 1-2 months before scheduled appointment. Patients also complete a survey at baseline and after standard of care colposcopy and an interview after standard of care colposcopy.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 21 to 65 years of age
* Had received an abnormal Pap smear result
* Scheduled colposcopy
* Able to communicate with ease in English or Spanish
* Have a cell phone with text (TXT) ability
* Competent to give consent

Exclusion Criteria:

* Are pregnant at the time of recruitment
* Display current evidence of positive invasive carcinoma of the cervix

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Patient Consent Rate | Up to 12 months
Study Completion Rate | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No